CLINICAL TRIAL: NCT01162642
Title: Green Tea Anticancer Mechanisms in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Diaz (Other)
Responsible Party: Sponsor-Investigator, Philip Diaz, M.D., Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007C0109
Record Dates: First submitted 2010-06-23; First posted 2010-07-14 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: Healthy moderately heavy smokers
MeSH Terms: conditions — Neoplasms | interventions — Tea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green Tea (Experimental): 4 cups daily of green tea for 6 weeks
  Interventions: Dietary Supplement: Green Tea
- No Green Tea (Placebo Comparator): 4 cups daily of placebo tea for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Green Tea — Green Tea 4 cups daily
  Arms: Green Tea
Other: Placebo — 4 cups placebo tea for 6 weeks
  Arms: No Green Tea

SUMMARY:
The purpose of this study is to determine whether green tea may lower the risk of certain cancers.

DETAILED DESCRIPTION:
Green tea contains phytochemicals, especially flavonoids. Phytochemicals are not absolutely required for normal functions, but may confer health benefits such as antioxidant actions. One can live without phytochemicals, but one may live longer and better with them. The phytochemicals in tea have been proposed to inhibit cancer onset via several different mechanisms. An obvious question is: Can anti-cancer actions of green tea be duplicated by black tea, which in the USA, is consumed more than green tea? The question remains unanswered, and will not be addressed by this project since many questions about green tea have not been answered yet. The contents of both type teas overlap in flavonoids, but green tea has more of the agents thought to be most effective. For example, some of the research cited below uses the flavonoid epigallocatechin gallate. Green tea has 5 times more of this flavonoid than black tea.

This study has two purposes. First, a case will be made that green tea may have several anti-cancer mechanisms, but this contention is not well confirmed by human intervention studies. This case will be made by addressing four questions. Second, justification will be given for the choice of mechanisms to be examined in this project's human intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 23-40 year old males and non-pregnant females, who are moderately heavy smokers (1-1.75 packs/day, > 2 years)

Exclusion Criteria:

* Habitual tea intake
* Habitual flavonoid supplementation
* Soy product intake over twice a week (soy is high in flavonoids).
* Pulmonary diseases
* Chronic or acute infection
* Admission of heavy alcohol intake (> 14 beers or drinks a week)
* Body mass index (BMI) > 30 (moderately overweight subjects will be taken)
* Abnormal EKG
* History of heart or other major health problems (ie arthritis, diabetes).
* Subjects with slightly high blood pressure will be eligible for the project, but more severe hypertension (>150/100)

Ages: 23 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Antioxidant effects of green tea versus placebo consumption. | Measured at post treatment
  Examine antioxidant effects of green tea versus placebo by measuring scavenging of free radicals; tea flavonoids; inflammatory cell secretion; endogenous antioxidant glutathione.

SECONDARY OUTCOMES:
Non-antioxidant, cancer-relevant effects of green tea consumption | Measured at pre-treatment and post treatment
  Examine non-antioxidant, cancer-relevant effects of green tea by measuring NF-kappaB inducing kinase; phosphorylation of cell signaling agents; tumor necrosis factor gene expression; lysyl oxidase enzyme; blockage of cancer cell proliferation.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Diaz, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States